CLINICAL TRIAL: NCT06762483
Title: Development and Validation of an Integrated Testing Strategy for Simultaneous Detection of ESR-1 and GBRCA Mutations Via Liquid Biopsy in HR+/HER2- Metastatic Breast Cancer (mBC) Patients, and the Creation of a Digital Gene Library to Support an Evidence-based Diagnostic Algorithm
Brief Title: Integrated Testing Strategy for Simultaneous Detection of ESR-1 and GBRCA Mutations Via Liquid Biopsy in HR+/HER2- Metastatic Breast Cancer (mBC) Patients,
Acronym: L2-268
Status: Recruiting | Type: Observational
Sponsor: European Institute of Oncology (Other)
Responsible Party: Sponsor
Other Study IDs: L2-268
Record Dates: First submitted 2024-12-31; First posted 2025-01-07 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2024-12

CONDITIONS: Breast Cancer, Metastatic
Keywords: HR+/HER2- BRCA
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Biospecimen Retention: Samples With DNA — blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- HR+/HER2- metastatic breast cancer (mBC) patients: breast

SUMMARY:
Development and validation of an integrated testing strategy for simultaneous detection of ESR-1 and gBRCA mutations via liquid biopsy in HR+/HER2- metastatic breast cancer (mBC) patients, and the creation of a digital gene library to support an evidence-based diagnostic algorithm

DETAILED DESCRIPTION:
Breast cancer is the most prevalent type of tumor and the primary cause of cancer-related deaths among women globally (1). Approximately two-thirds of these tumors express hormone receptors (HR) and lack HER2 overexpression and/or amplification (2). Throughout treatment, resistance frequently develops, with underlying mechanisms that remain largely undefined (3).

ELIGIBILITY:
Inclusion Criteria:

* Participants must have a confirmed diagnosis of estrogen receptor-positive (ER+) and/or progesterone receptor-positive (PgR+) breast cancer through histological and/or cytological examination by the local laboratory Participants must exhibit HER2-negative breast cancer

  1. or 2+). If IHC is 2+, a negative in situ hybridization (Fluorescent in situ hybridization (FISH), Chromogenic in situ hybridization (CISH), or Silver-enhanced in situ hybridization (SISH)) test is required by local laboratory testing.

     * Participants should be in an advanced or metastatic setting including both those prior to the initiation of treatment for metastatic disease and those who experienced progression following treatment with cyclin-dependent kinases (CDK)4/6 inhibitors. However, the primary tumor should be treated according to the standard of care.
     * Written informed consent must be signed and dated by the patient and the investigator prior to inclusion.

Exclusion Criteria:

* Unable to provide written informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible patients will be identified and enrolled in the study.
  * Blood sample collection and plasma purification Blood samples will be collected, and plasma will be purified following biobank procedures.
  * ESR1 and gBRCA liquid biopsy-based testing
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2024-12-20 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
the creation of a digital gene library to support an evidence-based diagnostic algorithm | 2 years
  Optimize the patient journey for individuals with metastatic breast cancer (mBC) by enhancing the care pathway and promoting access to testing for ESR1 and gBRCA mutations.

CONTACTS AND LOCATIONS:
Locations (1):
- European Institute of oncology, Milan, Italy, Italy